CLINICAL TRIAL: NCT06284291
Title: Use of Transcranial Magnetic Stimulation (TMS) as a Surrogate of Pathophysiology in Genetic Epilepsies
Brief Title: Transcranial Magnetic Stimulation (TMS) in Genetic Epilepsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Simona Balestrini, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TMSpath; RF-2021-12372804 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy; Genetic Disease
MeSH Terms: conditions — Epilepsy; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetic epilepsy (Experimental): Patients with epilepsies of genetic etiology
  Interventions: Diagnostic Test: transcranial magnetic stimulation (TMS)
- Patients with primary headache (Experimental): Patients with primary headache with non-migraine features
  Interventions: Diagnostic Test: transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Diagnostic Test: transcranial magnetic stimulation (TMS) — The STM9000 Standard-BI stimulator with 70 mm refrigerated butterfly stimulator (EB Neuro, Florence, Italy) controlled by Galileo Netbrain 9000 hardware and software (EB Neuro, Florence, Italy) is used. EMG data are recorded from the contralateral dorsal first interosseous muscle using gelled surface electrodes. EEG data are recorded by using the BE PLUS PRO Advanced EEG/EMG/EP amplifier (EB Neuro, Florence, Italy IT).

SUMMARY:
Transcranial magnetic stimulation (TMS) uses electromagnetic induction as an efficient, painless, non-invasive method to generate a suprathreshold current at the level of the encephalon, and provide in vivo measurements of cortical excitability and reactivity at the level of the motor cortex (TMS-EMG) or the entire cortical mantle (TMS-EEG). This study proposes TMS measurements as a diagnostic tool in patients to understand mechanisms of epileptogenesis related to genetic mutations, and prognostic to guide and monitor precision treatments.

ELIGIBILITY:
Inclusion Criteria:

* Children aged >3 years and adults
* Diagnosis of epilepsy with presumed or confirmed genetic etiology. Diagnosis of genetic epilepsy is made by next-generation sequencing (NGS) analysis
* or Diagnosis of primary (non-hemicranial) headache, in the absence of alterations on neuroimaging, and no known genetic condition
* Obtaining informed consent

Exclusion Criteria:

* Age <3 years
* Presence of contraindications to TMS: history of head or eye trauma with inclusion of metal fragments, cardiac pacemaker, arrhythmic heart disease, hearing implants, implantation of drug delivery devices, piercings or tattoos with metallic ink.
* Pregnancy status

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Resting motor threshold | 24 months
  Resting motor threshold (%MSO)
SICI | 24 months
  Short Interval intracortical inhibition (ratio)
ICF | 24 months
  Intracortical facilitation (ratio)
LICI | 24 months
  Long Interval Intracortical inhibition (ratio)
TEP amplitude | 24 months
  Amplitude of each component of the TMS-evoked potential (mV)
TEP latency | 24 months
  Latency of each component of the TMS-evoked potential (msec)

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Florence, Italy

IPD SHARING:
Plan to Share IPD: No